CLINICAL TRIAL: NCT05955885
Title: Effect of Over-the-counter Non-steroidal Anti-inflammatory Treatments on Cough Reflex Sensitivity in Subjects with Upper Respiratory Tract Infection
Brief Title: Effect of Over-the-counter NSAIDS on Cough Reflex Sensitivity in Patients with Upper Respiratory Tract Infections
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Reckitt Benckiser LLC (Industry)
Responsible Party: Principal Investigator, Stuart Mazzone, Professor in Neuroscience, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 25925
Record Dates: First submitted 2023-07-11; First posted 2023-07-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cough; Upper Respiratory Tract Infections
Keywords: Cough; Cough sensitivity; Urge to cough; Respiratory tract infection; Non-steroidal anti-inflammatory drug; Mechanism of disease
MeSH Terms: conditions — Cough; Respiratory Tract Infections | interventions — Benzydamine; Flurbiprofen

STUDY DESIGN:
Intervention Model Description: 120 participants will be randomised into four study arms, i.e. treatment with:
  1. flurbiprofen lozenge
  2. placebo lozenge
  3. flurbiprofen spray
  4. low dose flurbiprofen spray
  Regardless of which arm they are assigned to, each participant will undergo cough challenge testing to test cough sensitivity, fill out quality of life questionnaires, and have their nasal fluid, saliva and pharyngeal fluid sampled for inflammatory markers before and after the intervention.
Who Masked: Participant
Masking Description: The study will involve one-way blinding. Participants will be made aware prior to consenting that they will receive either flurbiprofen or a control intervention during the initial briefing and screening communications. However, they will not be told if the intervention they receive will contain flurbiprofen, a low dose of flurbiprofen, or no flurbiprofen. Blinding of the researchers to the identity of the treatment is difficult to achieve in practice given the physical characteristics of the interventions. Regardless of this, the researchers don't have any subjective role in quantifying the endpoint measures (patient-reported outcomes and cough sensitivity), minimising the risk of influencing the findings. For these reasons, the pragmatic approach of single blinding of the experiment is appropriate, acknowledging that this experiment is not designed to be a true clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Flurbiprofen Oral Lozenge (Experimental): 30 participants will be asked to suck one (1) flurbiprofen 8.75 mg honey and lemon lozenge (tradename: Strepfen) until dissolved.
  Interventions: Drug: Flurbiprofen Oral Lozenge
- Placebo lozenge (Placebo Comparator): 30 participants will be asked to suck one (1) non-medicated Difflam Soothing Drops + Immune Support Honey & Lemon flavour lozenge until dissolved.
  Interventions: Drug: Difflam
- Flurbiprofen 8.75 MG (Experimental): 30 participants will be asked to perform three (3) oral actuations (2.91 mg per actuation) of flurbiprofen 8.75mg spray.
  Interventions: Drug: Flurbiprofen 8.75 MG
- Low dose flurbiprofen spray (Other): 30 participants will be asked to perform one (1) oral actuation of flurbiprofen 8.75 mg spray, equivalent to a 2.91mg dosage. This will serve a a low dose control as there is no placebo spray available.
  Interventions: Drug: Flurbiprofen 8.75 MG

INTERVENTIONS:
Drug: Flurbiprofen Oral Lozenge — This commercially available, over-the-counter lozenge manufactured by Reckitt Benckiser contains flurbiprofen as the active ingredient and is registered for the short-term treatment of sore throat associated with upper respiratory tract infections in people over the age of 12 years.
  Other Names: Strepfen Intensive Lozenge - Honey and Lemon Flavour
  Arms: Flurbiprofen Oral Lozenge
Drug: Difflam — This is a non-medicated, control lozenge that is the same flavour as the experimental lozenge that is marketed to help soothe dry, tickly throats while supporting the body's immune health.
  Other Names: Difflam Soothing Drops + Immune Support Honey & Lemon Flavour
  Arms: Placebo lozenge
Drug: Flurbiprofen 8.75 MG — This commercially available, over-the-counter spray manufactured by Reckitt Benckiser contains flurbiprofen as the active ingredient and is registered for the short-term treatment of sore throat associated with upper respiratory tract infections in people over the age of 12 years. It requires 3 actuations of the spray to deliver the full 8.75 dose. Here, a low dose control can be delivered by only performing 1 actuation of the spray.
  Other Names: Strepfen Intensive Oromucosal Spray; Strepsils Intensive Oromucosal Spray
  Arms: Flurbiprofen 8.75 MG; Low dose flurbiprofen spray

SUMMARY:
The goal of this mechanism of disease study is to investigate the effect of flurbiprofen, a non-steroidal anti-inflammatory drug (NSAID), on the cough hypersensitivity associated with upper respiratory tract infections (URTI).

The main questions it aims to answer are:

* Q1: Does a single treatment with an approved therapeutic dose of flurbiprofen, an NSAID that prevents the production of prostaglandins, acutely reduce objective measures of cough hypersensitivity in participants with URTI?
* Q2: Is the effect of flurbiprofen on cough hypersensitivity in URTI related to participant subjective ratings of acute cough severity?
* Q3: Is the effect of flurbiprofen on cough hypersensitivity in URTI related to the levels of prostaglandins or other inflammatory markers measurable in upper airway secretions?

Participants will be asked to undergo cough challenge testing, complete quality of life questionnaires, and have their nasal fluid, saliva and pharyngeal secretions sampled before and after a single treatment with flurbiprofen in the form of a lozenge or spray. Participants in the comparator arms of the study will instead receive a placebo lozenge or low dose flurbiprofen spray.

DETAILED DESCRIPTION:
People with an Upper Respiratory Tract Infection (URTI), for example the common cold, often exhibit heightened sensitivity to stimuli that cause coughing. This heightened sensitivity is thought to contribute to the short-term excessive coughing that accompanies the infection. What causes the heightened sensitivity is not known but may involve inflammation in the throat.

HYPOTHESIS: The investigators hypothesise that in URTI prostaglandins may lead to cough hypersensitivity by either a direct or indirect action on cough nerve fibre endings in the larynx, lowering their activation threshold to cough stimuli.

OVERALL AIM: This study aims to investigate this hypothesis by assessing whether a single treatment with flurbiprofen, an existing over the counter anti-inflammatory drug (NSAID) medication contained in some 'cold and flu remedies' and used to relieve sore throat in URTI, reduces heightened cough sensitivity through a reduction in throat inflammation. The investigators will recruit 120 otherwise healthy male and female adults experiencing an URTI with acute cough for laboratory assessments lasting 5-6 hours.

OBJECTIVES: The primary objective is to assess whether flurbiprofen, in commercially available lozenge or spray formulations, reduces an individual's sensitivity to a cough evoking stimulus by assessing participant responsiveness to inhaled capsaicin. Capsaicin is the naturally occurring 'hot' component of chilli peppers and commonly used to investigate the cough reflex in humans.

The secondary objectives are to assess the effect of flurbiprofen on:

A. subjective measures of cough and urge-to-cough using questionnaires that assess Patient Reported Outcomes (PROs); and, B. the levels of chemical mediators of inflammation present in nasal secretions and saliva, to investigate flurbiprofen's potential mechanism of action.

METHOD: The investigators will test the hypothesis by measuring in participants their cough thresholds, subjective experiences with cough and urge-to-cough, and levels of airway prostaglandins and other inflammatory mediators, before and after a single treatment of flurbiprofen, which blocks the production of prostaglandins.

ELIGIBILITY:
Inclusion Criteria:

* An onset of any 2 URTI symptoms in past 3-5 days, such as a sore throat, fever, coughing, coughing up phlegm, sneezing, and runny nose;
* A current cough or urge-to-cough rated at least 5 in severity and/or ranking cough as subject's most bothersome symptom on Cold Symptoms Questionnaire (CSQ);
* A feeling of sickness interfering with their daily life, rated as at least mildly;
* A cough consistent with acute cough - i.e., cough onset with URTI and not ongoing, chronic cough;
* Written informed consent and a willingness and ability to comply with the study protocol.

Exclusion Criteria:

* A pre-existing chronic lung disease (asthma, COPD, chronic bronchitis etc), to exclude these as causes for cough;
* The use of inhaled or systemic steroids / broncho-active medication, ACE inhibitors, oral or inhaled antihistamines, opiates, gabapentin, tricyclic antidepressants (current or within the past 3 months), as these will alter airway inflammatory profiles and/ or cough sensitivity;
* A current cigarette or marijuana smoker/vaper, recreational drug user, or have given up smoking/vaping within the last 12 months, or a former smoker with greater than 20 pack-years, alter airway inflammatory profiles and/ or cough sensitivity;
* Pre-existing chronic cough (cough persisting for more than 8 weeks): unexplained chronic cough (UCC) or refractory chronic cough (RCC) associated with or without a pre-existing condition (GERD, rhinitis, etc), as we are studying acute cough;
* Prior experience of an allergic or bad reaction to capsaicin or chilli (which is rare);
* Prior experience an allergic or bad reaction to a non-steroidal anti-inflammatory drug (NSAID) such as ibuprofen;
* Ongoing or history of stomach ulcer, impaired kidney or liver function, or heart failure;
* Pregnancy, lactation or actively trying to become pregnant;
* Currently taking other products with flurbiprofen, aspirin or other anti-inflammatory medicines;
* Evidence of COVID-19 positivity, either during the COVID Rapid Antigen Test administered on the day of assessment or have informed us that they have become positive in the 24-48 hours after the testing session (i.e., participants who were likely positive during assessment but under the detection threshold);
* Participants who cannot provide informed voluntary consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in objective measures of cough sensitivity | Cough challenge testing will be performed at baseline and 3 hours after intervention.
  Participants' cough sensitivity thresholds will be measured by inhaled cough challenge testing. This involves participants inhaling single breaths of increasing concentrations of a tussigenic stimulus (capsaicin; (active component of hot chili peppers) as well as saline control to determine threshold doses that elicit an urge to cough, two coughs (C2) and five coughs (C5). The principal endpoint is measured as the change in capsaicin concentration needed to elicit cough responses and the unit of measure is micromolar.

SECONDARY OUTCOMES:
Change in Cold Symptoms Questionnaire (CSQ) score | Participant self-reports using the Cold Symptoms Questionnaire at baseline and every 30 min after invention until 3 hours has elapsed.
  Participants will be asked to self-report on their cold symptom severity using the Cold Symptoms Questionnaire. Each item requires rating on a 10-point Likert scale from 1 to 10. A higher score indicates a worse outcome. The principal endpoint is measured as the change in Cold Symptoms Questionnaire score and the unit of measure is points.
Change in levels of inflammatory markers in nasal fluid samples | Nasal fluid samples will be taken at baseline and at 3 hours post-intervention.
  Samples of nasal fluid will be taken from participants and levels of inflammatory markers such as prostaglandins will be measured using liquid chromatography-mass spectroscopy. The principle endpoint is measured as change in levels and the unit of measure is points. A higher score indicates a better outcome.
Change in levels of inflammatory markers in saliva samples | Saliva samples will be taken at baseline and at 3 hours post-intervention.
  Samples of saliva will be taken from participants and levels of inflammatory markers such as prostaglandins will be measured using liquid chromatography-mass spectroscopy. The principle endpoint is measured as change in levels and the unit of measure is points. A higher score indicates a better outcome.
Change in levels of inflammatory markers in pharyngeal lavage samples | Pharyngeal lavage samples will be taken at baseline and at 3 hours post-intervention.
  Samples of pharyngeal fluid and tissue will be collected from a lavage and levels of inflammatory markers such as prostaglandins will be measured using liquid chromatography-mass spectroscopy. The principle endpoint is measured as change in levels and the unit of measure is points. A higher score indicates a better outcome.
Patients' Global Impression of Change score | Participants self-report using the Patients' Global Impression of Change score at 3 hours post-intervention.
  Participants will self-report on their overall impression of whether the intervention they received resulted in any perceivable changes in their coughing/urge-to-cough. This questionnaire contains mixed items, including items that require rating of degree of change of symptoms on a 10 point Likert scale. The principal endpoint is the score for each item and the unit of measure is points.A higher score indicates a worse outocme.

OTHER OUTCOMES:
Leicester Cough Questionnaire - Acute score | Participants self-report using the Leicester Cough Questionnaire at baseline.
  Participants will be asked to self-report on the impact of cough on their quality of life to enable a measurement of how severe their cough is at baseline. Each item requires a rating on a 7-point Likert scale from 1 to 7 and is related to the impact of cough in one of three domains (physical, psychological social). The Leicester Cough Questionnaire is scored by averaging the ratings in each domain and then adding the average domain scores (range 3-21). A higher score indicates a better outcome. The principal endpoint is measured as the overall Leicester Cough Questionnaire score and the unit of measure is points.
Optional: Acute Cough Scale (ACS) score | Participants self-report using the Acute Cough Scale at baseline.
  Inclusion of this scale is exploratory and participants may choose to do it. It is new, alternative scale to a Visual Analogue Scale that enables the respondent to describe their cough in a more detailed fashion through 13 items that capture specific dimensions of cough and using a 6 point Likert scale from 0 to 5 with cues given at each grade. The principle endpoint is measured as total score and the unit of measure is points. A higher score indicates a greater severity of cough and disturbance to daily well-being, i.e. worse outcome.
Optional: 8-item Quality of Life General (QGEN-8) survey | Participants self-report using the 8-item Quality of Life General survey at baseline.
  Inclusion of this scale is exploratory and participants may choose to do it. It is new survey that condenses the numerous items measuring functional health and well-being in other, lengthy health-related quality of life surveys into an 8-item survey that reduces the time and effort burden on survey respondents. It also extends the measurement range to reduce ceiling effects commonly noted in the functioning and feeling domains. The principle endpoint is measured as total score and the unit of measure is points. A higher score indicates a greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mazzone, PhD, Principal Investigator — University of Melbourne
Locations (1):
- University of Melbourne, Carlton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazzone SB, Farrell MJ. Heterogeneity of cough neurobiology: Clinical implications. Pulm Pharmacol Ther. 2019 Apr;55:62-66. doi: 10.1016/j.pupt.2019.02.002. Epub 2019 Feb 11. PMID 30763726
- [Background] Farrell MJ, Mazzone SB. Are neural pathways processing airway inputs sensitized in patients with cough hypersensitivity? Pulm Pharmacol Ther. 2019 Aug;57:101806. doi: 10.1016/j.pupt.2019.101806. Epub 2019 May 15. PMID 31100512
- [Background] Dicpinigaitis PV. Effect of viral upper respiratory tract infection on cough reflex sensitivity. J Thorac Dis. 2014 Oct;6(Suppl 7):S708-11. doi: 10.3978/j.issn.2072-1439.2013.12.02. PMID 25383204
- [Background] Driessen AK, McGovern AE, Narula M, Yang SK, Keller JA, Farrell MJ, Mazzone SB. Central mechanisms of airway sensation and cough hypersensitivity. Pulm Pharmacol Ther. 2017 Dec;47:9-15. doi: 10.1016/j.pupt.2017.01.010. Epub 2017 Jan 27. PMID 28137663
- [Background] Renner B, Mueller CA, Shephard A. Environmental and non-infectious factors in the aetiology of pharyngitis (sore throat). Inflamm Res. 2012 Oct;61(10):1041-52. doi: 10.1007/s00011-012-0540-9. Epub 2012 Aug 14. PMID 22890476
- [Background] Lambkin-Williams R, Mann A, Shephard A. Inhibition of viral and bacterial trigger-stimulated prostaglandin E2 by a throat lozenge containing flurbiprofen: An in vitro study using a human respiratory epithelial cell line. SAGE Open Med. 2020 Sep 24;8:2050312120960568. doi: 10.1177/2050312120960568. eCollection 2020. PMID 33029351
- [Background] Schachtel BP, Homan HD, Gibb IA, Christian J. Demonstration of dose response of flurbiprofen lozenges with the sore throat pain model. Clin Pharmacol Ther. 2002 May;71(5):375-80. doi: 10.1067/mcp.2002.124079. PMID 12011823
- [Background] Schachtel B, Aspley S, Shephard A, Shea T, Smith G, Sanner K, Savino L, Rezuke J, Schachtel E. Onset of action of a lozenge containing flurbiprofen 8.75 mg: a randomized, double-blind, placebo-controlled trial with a new method for measuring onset of analgesic activity. Pain. 2014 Feb;155(2):422-428. doi: 10.1016/j.pain.2013.11.001. Epub 2013 Nov 12. PMID 24231654